CLINICAL TRIAL: NCT06518785
Title: Ultrasound Neuromodulation of the Brain for Alcohol Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 24-41883
Record Dates: First submitted 2024-07-08; First posted 2024-07-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use Disorder
Keywords: Substance Use Disorder; Low-Intensity Focused Ultrasound; Transcranial Focused Ultrasound; Neuromodulation
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: This is a single-center, double-blind, controlled, randomized, complete block, 2-period crossover pilot trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the objectives of the study, the identity of LIFU treatments will not be known to research staff performing the data analysis or participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- VS LIFU/ VPL LIFU (Experimental): Participants will be assigned to receive VS LIFU during the first LIFU treatment session.
  Interventions: Device: Low Intensity Focused Ultrasound
- VPL LIFU/VS LIFU (Active Comparator): Participants will be assigned to receive VPL LIFU during the first LIFU treatment session.
  Interventions: Device: Low Intensity Focused Ultrasound

INTERVENTIONS:
Device: Low Intensity Focused Ultrasound — An inhibitory LIFU protocol that allows suppression of neuronal activity in the basal ganglia and thalamus will be used.
  Other Names: LIFU

SUMMARY:
This study aims to examine the effects of Low-Intensity Focused Ultrasound (LIFU) on brain activity in patients with alcohol use disorder.

DETAILED DESCRIPTION:
This is a single-center, double-blind, controlled, randomized, complete block, 2-period crossover pilot trial. The study will assess target engagement of the ventral striatum after LIFU in patients with alcohol use disorder using resting state and task-based functional magnetic resonance imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. Documentation of an AUD diagnosis per DSM-5 criteria as evidenced by problematic pattern of alcohol use leading to clinically significant impairment or distress, as manifested by at least two of the DSM-5 criteria, occurring within a 12-month period.
3. Be willing to undergo a brain MRI and follow study protocol.

Exclusion Criteria:

1. Pregnant or breastfeeding.
2. Presence of a condition or abnormality that would compromise the safety of the patient or the quality of the data.
3. Non-English speaking.
4. Other investigational AUD treatments.
5. Primary psychosis, Bipolar I, or severe personality disorder.
6. Active suicidality or history of suicide attempt in the past 5 years.
7. Cognitive impairment (MoCA <24)
8. Significant medical or neurological disease, or life expectancy <12 mos.
9. Significant brain abnormality on brain imaging.
10. Any MRI exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of LIFU-related adverse events. | Through study completion, an average of 5 weeks
  This will be assessed through monitoring for adverse events (AE) throughout the study.
Reward network activity in response to alcohol cues. | 3 visits over 3 weeks
  Reward network activity in response to alcohol vs. neutral cues before and after LIFU will be assessed using fMRI.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Moussawi, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarica C, Nankoo JF, Fomenko A, Grippe TC, Yamamoto K, Samuel N, Milano V, Vetkas A, Darmani G, Cizmeci MN, Lozano AM, Chen R. Human Studies of Transcranial Ultrasound neuromodulation: A systematic review of effectiveness and safety. Brain Stimul. 2022 May-Jun;15(3):737-746. doi: 10.1016/j.brs.2022.05.002. Epub 2022 May 6. PMID 35533835
- [Background] Legon W, Adams S, Bansal P, Patel PD, Hobbs L, Ai L, Mueller JK, Meekins G, Gillick BT. A retrospective qualitative report of symptoms and safety from transcranial focused ultrasound for neuromodulation in humans. Sci Rep. 2020 Mar 27;10(1):5573. doi: 10.1038/s41598-020-62265-8. PMID 32221350
- [Background] Stern JM, Spivak NM, Becerra SA, Kuhn TP, Korb AS, Kronemyer D, Khanlou N, Reyes SD, Monti MM, Schnakers C, Walshaw P, Keselman I, Cohen MS, Yong W, Fried I, Jordan SE, Schafer ME, Engel J Jr, Bystritsky A. Safety of focused ultrasound neuromodulation in humans with temporal lobe epilepsy. Brain Stimul. 2021 Jul-Aug;14(4):1022-1031. doi: 10.1016/j.brs.2021.06.003. Epub 2021 Jun 23. PMID 34198105
- [Background] Mahoney JJ, Haut MW, Carpenter J, Ranjan M, Thompson-Lake DGY, Marton JL, Zheng W, Berry JH, Tirumalai P, Mears A, D'Haese P, Finomore VS, Hodder SL, Rezai AR. Low-intensity focused ultrasound targeting the nucleus accumbens as a potential treatment for substance use disorder: safety and feasibility clinical trial. Front Psychiatry. 2023 Sep 15;14:1211566. doi: 10.3389/fpsyt.2023.1211566. eCollection 2023. PMID 37779628
- [Background] Martin E, Aubry JF, Schafer M, Verhagen L, Treeby B, Pauly KB. ITRUSST consensus on standardised reporting for transcranial ultrasound stimulation. Brain Stimul. 2024 May-Jun;17(3):607-615. doi: 10.1016/j.brs.2024.04.013. Epub 2024 Apr 25. PMID 38670224